CLINICAL TRIAL: NCT03234959
Title: CareToy: a Smart System for Early Home-based Intervention in Infants at High Risk for Cerebral Palsy
Brief Title: CareToy Early Intervention in Infants at Risk for Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RF-2013-02358095 CareToy
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy
Keywords: Early Intervention; Cerebral Palsy; CareToy Intervention; Infant Massage; Information Communication Technology
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CareToy Intervention (Experimental): Infants will perform individualized goal-directed activities for 30-45 minutes per day with CT system, while continuing SC. The CT training will be monitored and modified remotely by clinical staff, according to infants' developmental needs, abilities and progresses. It will last 8 wks.
  Interventions: Device: CareToy intervention
- Infant Massage (Active Comparator): Infants and their caregivers will perform 4-5 sessions (around 1 hour every 2 weeks) of Infant massage conducted by an expert child therapist. The therapist will instruct the parent in the baby's massage and provide advises on promoting development. Parents will be invited to perform infant massage five days a week, for 8 weeks. Parent will take a diary in which will record the frequency of the IM.
  Interventions: Other: Infant Massage

INTERVENTIONS:
Device: CareToy intervention — Infants will perform goal directed activities inside the CareToy System
  Other Names: CT
  Arms: CareToy Intervention
Other: Infant Massage — Infants will received IM by their parents
  Other Names: IM
  Arms: Infant Massage

SUMMARY:
Cerebral Palsy (CP), due to pre-perinatal brain lesions, is a main cause of childhood disabilities with high cost for individuals and society. Early Intervention (EI), if intensive enough but affordable by patients, family and health services can improve its outcome. A recent Cochrane review indicates the positive effects of Infant Massage (IM) in gross and fine motor skills, visual development and parent infants interaction in preterm infants. Recently, a new technological tool, called CareToy has been developed as a tele-rehabilitation tool for delivering at home EI. The effects of CT training on neurodevelopmental outcome have been recently tested in a sample of low-risk preterm infants with very promising results. The aim of the project is to provide evidence, by a RCT, of the efficacy of CareToy (CT) training versus Infant Massage, in a sample of 45 infants aged 3-12 months (or with motor competencies from initial head control to unstable sitting position) at high risk for CP according to strict clinical and neuroradiological signs. Enrolled infants will be randomized in 2 groups: CareToy and Infant Massage. Infants allocated in CT group will perform a training with CT while the others will perform infant massage. Both trainings will be carried out at home by parents with the monitoring of the therapists. Both interventions will last 8 weeks. All enrolled infants will be evaluated at baseline (T0),9 wks after the CT/IM (T1), 9 wks after T1 (T2) and at 18 months of post term age (T3). Infant Motor Profile will be the primary outcome measure.

DETAILED DESCRIPTION:
The eligibility of infants, i.e. infants who meet the criteria for inclusion and exclusion (i.e infants at high-risk for CP) will be evaluated by the Neonatology team and the recruitment will be done after discharge from Neonatal Intensive Care Unit (NICU) during the follow up performed by infants previously enrolled in the first observational phase (aimed to identify infants at high risk for CP) and will begin with the signing of the participation agreement by the parents. The study is designed as randomized clinical trial. Recruited infants will be randomized in two groups: CareToy intervention vs Infant Massage. All infants will perform the home based and family centered early intervention according to their allocation group for 8 weeks. Before (T0), after the intervention period (T1) and in follow up (at T2, 8 wks after T1 and at 18 mths of post term age) all infants will be evaluated with standardized scales and questionnaires in order to evaluate the effects of EI on motor, cognitive and visual development and parent-infant interaction. Moreover the sleep organization, before and after the intervention, will be studied using actigraphs. The sample size has been calculated on the basis of the primary outcome measure (Infant Motor Profile).

ELIGIBILITY:
Inclusion Criteria:

* i) abnormal neurological signs (i.e. neurological signs at the Hammersmith Infant Neurological Assessment -HINE- and according to Prechtl's Assessment GMA) at 2-4 mts post term age
* ii) neuroimaging evidence of brain lesion indicated by MRI performed around the term age (4-6 wks post term)
* iii) achieved predefined motor development scores assessed by Ages and Stages Questionnaire-3
* iv) informed consent agreement

Exclusion Criteria:

* i) Drug resistant seizures,
* ii) Severe sensory deficits (blindness or deafness)
* iii) Progressive neurological disorders
* iv) Malformation of CNS

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Changes in Infant Motor Profile (IMP) | Baseline (i.e within 1 week before the beginning of study, T0); within 1 week after the CT/IM period (T1); 8 weeks after the end of CT/IM periods (T2); at 18 mths of post term age (T3)
  It is a video-based and qualitative assessment of motor behaviour in infancy, applicable in preterm and at term infants aged 3 to 18 months. It consists of 80 items addressed to explore the child's motor abilities and to evaluate motor behaviour.

SECONDARY OUTCOMES:
Changes in Peabody Developmental Motor Scales Second Edition (PDMS-2) | Baseline (i.e within 1 week before the beginning of study, T0); within 1 week after the CT/IM period (T1); 8 weeks after the end of CT/IM periods (T2), at 18 mths of post term age (T3)
  PDMS-2 is composed of six subtests that measure interrelated abilities in early motor development. It was designed to assess gross and fine motor skills in children from birth through five years of age.
Changes in Teller Acuity Cards | Baseline (i.e within 1 week before the beginning of study, T0); within 1 week after the CT/IM period (T1); 8 weeks after the end of CT/IM periods (T2); at 18 mths of post term age (T3)
  Teller Acuity Cards are used to evaluate visual acuity in infants and children. It is based on judgement of the infant attention to a series of cards showing stripes of different widths. This tool allows rapid assessment of resolution (grating) visual acuity in infants and young children.
Changes in Bayley Cognitive subscale (BSID-III) | Baseline (i.e within 1 week before the beginning of study, T0); at 18 mths of post term age (T3)
  This scale is sensitive in detecting differences between a normative sample and children at risk for delayed development, such as premature infants. Bayley III is appropriate for administration to children between the ages of 1 month and 42 months.
Changes in Care-Index | Baseline (i.e within 1 week before the beginning of study, T0); within 1 week after the CT/IM period (T1); 8 weeks after the end of CT/IM periods (T2); at 18 mths of post term age (T3)
  It assesses caregiver-infant interaction from birth to about two years of age based on a short, videotaped play interaction of 3-5 minutes. The measure assesses caregivers on three scales: sensitivity, control and unresponsiveness. There are also four scales for infants: cooperativeness, compulsivity, difficultness, and passivity.
Changes in sleep organization | Baseline (i.e within 1 week before the beginning of study, T0); within 1 week after the end of the CT/IM period (T1)
  It is simpler and less invasive survey instrument for the objective assessment of the sleep, which allows for prolonged monitoring (from days to months). It uses acceleration sensors, the size of a watch, usually worn on the wrist the non-dominant hand. Dedicated algorithms have been developed to the identification of sleep in pediatric populations.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Tirrenia, Tuscany, Italy

REFERENCES:
- [Background] Sgandurra G, Beani E, Giampietri M, Rizzi R, Cioni G; CareToy-R Consortium. Early intervention at home in infants with congenital brain lesion with CareToy revised: a RCT protocol. BMC Pediatr. 2018 Sep 5;18(1):295. doi: 10.1186/s12887-018-1264-y. PMID 30185165
- [Derived] Franchi De' Cavalieri M, Filogna S, Martini G, Beani E, Maselli M, Cianchetti M, Dubbini N, Cioni G, Sgandurra G; CareToy-R Consortium. Wearable accelerometers for measuring and monitoring the motor behaviour of infants with brain damage during CareToy-Revised training. J Neuroeng Rehabil. 2023 May 6;20(1):62. doi: 10.1186/s12984-023-01182-z. PMID 37149595
- [Derived] Menici V, Antonelli C, Beani E, Mattiola A, Giampietri M, Martini G, Rizzi R, Cecchi A, Cioni ML, Cioni G, Sgandurra G; Caretoy-R Consortium. Feasibility of Early Intervention Through Home-Based and Parent-Delivered Infant Massage in Infants at High Risk for Cerebral Palsy. Front Pediatr. 2021 Jul 19;9:673956. doi: 10.3389/fped.2021.673956. eCollection 2021. PMID 34350144
- [Derived] Rizzi R, Menici V, Cioni ML, Cecchi A, Barzacchi V, Beani E, Giampietri M, Cioni G, Sgandurra G; Clinical CareToy-R Consortium. Concurrent and predictive validity of the infant motor profile in infants at risk of neurodevelopmental disorders. BMC Pediatr. 2021 Feb 6;21(1):68. doi: 10.1186/s12887-021-02522-5. PMID 33549070